CLINICAL TRIAL: NCT02204293
Title: Study Protocol for a Multi-Centre, Placebo-Controlled Phase II Study of Canakinumab for the Treatment of Adult-onset Still's Disease (AOSD) Including an Open-label Long Term Extension
Brief Title: Canakinumab for Treatment of Adult-onset Still's Disease
Acronym: CONSIDER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment issues due to marketing authorization of study drug
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Eugen Feist, Prof. Dr Eugen Feist, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CACZ885GDE01T; 2011-001027-20 (EudraCT Number)
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Adult-Onset Still´s Disease
Keywords: Adult-Onset Still´s Disease; Canakinumab; Joint involvement; AOSD
MeSH Terms: interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canakinumab (Experimental): Participants received canakinumab 4 mg/kg up to a maximum of 300 mg subcutaneous (SC) injection, once in morning on Day 0, Weeks 4, 8, and 12 in Part I of the core study. Participants with response (change in DAS score > 1.2 at Week 12) continued to receive same dose of canakinumab in Part II for Weeks 12, 16, and 20. Participants who had remission (change in DAS score > 1.2 and no signs of systemic activity for adult-onset Still's disease at Week 20) entered Long-term extension (LTE) phase and received same dose of canakinumab at Weeks 24 and 28, which was down titrated to 2 mg/kg if applicable from Week 28 up to Month 27.
  Interventions: Drug: Canakinumab
- Placebo (Placebo Comparator): Participants received placebo, SC injection, once in morning on Day 0, Weeks 4, 8, and 12 in Part I of the core study. Participants with response (change in DAS score > 1.2 at Week 12) continued to receive placebo at Weeks 12, 16, and 20. Non-responders (who had change in DAS score ≤ 1.2) were unblinded to receive canakinumab 4 mg/kg (up to 300 mg maximum), SC injection, at Weeks 12, 16, and 20. Participants who had remission (change in DAS score > 1.2 and no signs of systemic activity for adult-onset Still's disease at Week 20) entered Long-term extension (LTE) phase and received same dose of canakinumab at Weeks 24 and 28, which was down titrated to 2 mg/kg if applicable from Week 28 up to Month 27.
  Interventions: Drug: Canakinumab; Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab — Canakinumab, single-dose 4 mg/kg up to 300 mg administered subcutaneously.
  Other Names: Ilaris
Drug: Placebo — Matching placebo administered subcutaneously.
  Arms: Placebo

SUMMARY:
The purpose of this trial is to investigate the efficacy of the treatment with canakinumab in participants with Adult-onset Still's Disease (AOSD) and active joint involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed consent from the participant to take part in the study
2. Men and women aged ≥ 18 years and ≤ 75 years
3. Fulfilment of AOSD classification criteria (according to Yamaguchi et al, J. Rheumatology, 1992)
4. Disease activity based on Disease Activity Score 28 (DAS28) of ≥3.2 at screening
5. At least 4 painful and 4 swollen joints at screening and baseline (of the 28 joints according to DAS28)
6. If undergoing treatment with non-steroidal anti-inflammatory drugs (NSAIDs), stable dose for at least 4 weeks prior to randomisation
7. If undergoing treatment with glucocorticoids, stable dose of ≤10 milligrams per day (mg/day) (prednisolone or equivalent) for at least 4 weeks prior to randomisation
8. If undergoing treatment with conventional disease-modifying anti-rheumatic drugs (DMARD), stable dose for at least 3 months prior to randomisation
9. Normalisation period for biological DMARDS (anakinra 1 week, etanercept 1 month, adalimumab and certolizumab 2 months, infliximab, golimumab, abatacept and tocilizumab 3 months, rituximab 9 months, canakinumab 6 months) prior to randomisation
10. In participants of reproductive age, use of an effective method of contraception as well as negative pregnancy test prior to the study commencing.

Exclusion Criteria:

1. Previous treatment with the study drug with repeated administration of canakinumab
2. Intraarticular or intravenous administration of glucocorticoids within 4 weeks prior to the baseline or use of narcotic analgesics except for analgesics permitted within the framework of the investigation (codeine and tramadol)
3. Presence of another, serious chronic-inflammatory disease
4. Positive hepatitis B antigen (HBsAg), hepatitis C antibodies and/or human immunodeficiency virus (HIV) antibodies.
5. Presence of a relevant, active infection or other diseases, which entail a tendency towards infection
6. Positive screening for latent tuberculosis, in accordance with usual local practice
7. Raised liver count (raised bilirubin; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3-fold the normal range)
8. Serum-creatinine concentration >1.5 milligrams per deciliter (mg/dL)
9. Inadequate haematological findings (hemoglobin [Hb] ≤ 10 grams per deciliter (g/dL), neutrophils ≤2,500/microliter (µl) and thrombocytes ≤100,000/µl)
10. Simultaneous participation in any other interventional clinical study within the last 30 days preceding the commencement of the study
11. History of neoplasia with the exception of a curatively treated non-melanoma skin tumour or carcinoma of the cervix treated in situ without any indication of recurrence within the last 10 years
12. Relevant cardiac or pulmonary disorders
13. Severe intercurrent neurological or psychiatric disorders
14. Macrophage activation syndrome (MAS) as part of previous treatment with IL-1 blockade (e.g. anakinra, rilonacept)
15. Vaccination with a live vaccine within 3 months before the baseline
16. Alcohol or drug abuse in the past 12 months
17. ≥400 milliliter (mL) donation of blood or loss up to 8 weeks before the baseline
18. Pregnancy or breast-feeding
19. Commitment of the patient to an institution at the direction of an authority or court

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-06-21 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugen Feist, Prof. Dr., Principal Investigator — Charité University Berlin Germany
Locations (14):
- Germany (14):
  - Charité Campus Mitte, Berlin
  - Immanuel Krankenhaus Berlin, Berlin
  - Med. Klinik I für Innere Medizin Köln, Cologne
  - Universität Erlangen, Erlangen
  - Kliniken Essen-Süd/Krankenhaus St. Josef, Essen
  - Universitätsklinikum der J.W. Goethe-Universität Frankfurt, Frankfurt A. M.
  - Asklepios Klinikum Hamburg Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätskrankenhaus Schleswig Holstein, Kiel
  - Klinikum der Universität München, München
  - Klinikum Südstadt Rostock, Rostock
  - Universitätsklinikum Tübingen, Tübingen
  - Fachkrankenhaus, Vogelsang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nirmala N, Brachat A, Feist E, Blank N, Specker C, Witt M, Zernicke J, Martini A, Junge G. Gene-expression analysis of adult-onset Still's disease and systemic juvenile idiopathic arthritis is consistent with a continuum of a single disease entity. Pediatr Rheumatol Online J. 2015 Nov 20;13:50. doi: 10.1186/s12969-015-0047-3. PMID 26589963
- See also: Related Info — http://ard.bmj.com/content/early/2020/05/13/annrheumdis-2020-217155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with adult-onset Still's disease (AOSD) took part in the study from June 21, 2012 to May 5, 2018 at 14 investigative sites located in Germany to participate in two double-blind parts - Part I (Up to Week 12) and Part II (Up to Week 24) and one open-label Long-Term Extension (LTE) phase (Up to Month 27).
Pre-assignment Details: A total of 36 participants entered in Part I to receive canakinumab/placebo. Out of 31, 5 participants from canakinumab arm, and 3 from placebo arm did not enter Part II, 23 participants entered Part II and received canakinumab or placebo up to Week 24. 7 participants who achieved clinical remission entered LTE Phase to receive canakinumab.
Groups:
- Core Study Part I: Canakinumab: Participants received canakinumab 4 mg/kg up to 300 mg maximum, subcutaneous (SC) injection, once in morning at Baseline (Day 0), Weeks 4, 8, and 12.
- Core Study Part I: Placebo: Participants received placebo, SC injection, once in morning at Baseline (Day 0), Weeks 4, 8, and 12.
- Core Study Part II: Canakinumab Responders: Participants with response (change in DAS score > 1.2 at Week 12) continued to receive canakinumab 4 mg/kg up to 300 mg maximum, SC injection, once in the morning for Weeks 12, 16, and 20.
- Core Study Part II: Placebo Responders: Participants with response (change in DAS score > 1.2 at Week 12) continued to receive placebo, SC injection, once in morning for Weeks 12, 16, and 20.
- Core Study Part II: Placebo Non-responders: Placebo Non-responders (change in DAS score ≤ 1.2 at Week 12) who switched to canakinumab were unblinded to receive canakinumab 4 mg/kg up to 300 mg maximum, SC injection, once in the morning at Weeks 12, 16, and 20.
- LTE Phase: Canakinumab: Participants with remission (change in DAS score > 1.2 and no signs of systemic activity for adult-onset Still's disease at Week 20) received canakinumab 4 mg/kg up to 300 mg maximum, SC injection at Weeks 24 and 28, which was down titrated to 2 mg/kg up to 150 mg maximum if applicable after Week 28 up to Month 27 (Week 117).
Period: Core Study Part I
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo | Core Study Part II: Canakinumab Responders | Core Study Part II: Placebo Responders | Core Study Part II: Placebo Non-responders | LTE Phase: Canakinumab
Started | 19 | 17 | 0 | 0 | 0 | 0
Intention-to-treat Population | 18 (One participant left the study before treatment was started.) | 17 | 0 | 0 | 0 | 0
Safety Population | 20 (2 participants from placebo arm received canakinumab at Week 4, included in Safety population.) | 15 | 0 | 0 | 0 | 0
Completed | 17 | 14 | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Met one or more exclusion criteria | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 3 | 0 | 0 | 0 | 0
Period: Core Study Part 2
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo | Core Study Part II: Canakinumab Responders | Core Study Part II: Placebo Responders | Core Study Part II: Placebo Non-responders | LTE Phase: Canakinumab
Started | 0 (Participants who achieved response at Week 12, entered Part II.) | 0 | 12 (Participants who achieved response at Week 12, entered Part II.) | 4 | 7 | 0
Safety Population | 0 | 0 | 14 (Included 2 participants from placebo arm who received canakinumab at Week 4.) | 2 | 7 | 0
Completed | 0 | 0 | 12 | 4 | 7 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: LTE Phase
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo | Core Study Part II: Canakinumab Responders | Core Study Part II: Placebo Responders | Core Study Part II: Placebo Non-responders | LTE Phase: Canakinumab
Started (Participants who achieved remission entered LTE Phase.) | 0 | 0 | 0 | 0 | 0 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 7
Not completed — Study Suspended | 0 | 0 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all participants who did not violate any of the following inclusion criteria: diagnosis of adult-onset Still's disease and disease activity based on DAS28 score of ≥ 3.2 at Screening.
Groups:
- Total: Total of all reporting groups
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.06 (13.2) | 40.53 (13.2) | 40.79 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 8 | 4 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Core Study Part I: Percentage of Responders as Assessed by Disease Activity Score 28 Joints (DAS28) Score at Week 12
Description: Responders included participants with change in disease activity score based on 28 joint counts and ESR (DAS28) score > 1.2. The DAS28 score index is a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, patient global assessment of disease activity score, and the erythrocyte sedimentation rate (ESR) value. Total score ranged between 0-10. A DAS28-ESR score of 5.1 or above = high disease activity, a value between 3.2 and 5.1 = moderate disease activity and value between 2.6 and 3.2 = low disease activity, value < 2.6 = disease remission.
Time Frame: Week 12
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
percentage of participants | 66.7 [43.1 to 85.2] | 41.2 [20.1 to 65.0]
Statistical Analysis 1: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 0.1811, Fisher Exact

2. Secondary Outcome: Core Study Part I: Change From Baseline (CFB) in Disease Activity Score 28 Joints Erythrocyte Sedimentation Rate (DAS28 [ESR]) Score
Description: The DAS28 index is a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, patient global assessment of disease activity score, and ESR value.Total score ranged between 0-10. A DAS28-ESR score of 5.1 or above = high disease activity, a value between 3.2 and 5.1 = moderate disease activity and value between 2.6 and 3.2 = low disease activity, value < 2.6 = disease remission. A positive change in score indicates worsening, and a negative change indicates improvement. Least squares (LS) mean was calculated by mixed linear model for repeated measures (MMRM) analyses.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: ITT population included all participants who did not violate any of the following inclusion criteria: diagnosis of adult-onset Still's disease and disease activity based on DAS28 score of ≥ 3.2 at Screening. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
score on a scale
  Baseline | 5.37 [4.7 to 6.0] | 5.3 [4.6 to 6.0]
  CFB at Week 4: number analyzed (Participants) | 16 | 14
  CFB at Week 4 | 3.56 [2.9 to 4.3] | 4.27 [3.5 to 5.0]
  CFB at Week 8: number analyzed (Participants) | 16 | 12
  CFB at Week 8 | 2.86 [2.2 to 3.6] | 3.92 [3.1 to 4.7]
  CFB at Week 12: number analyzed (Participants) | 16 | 14
  CFB at Week 12 | 3.1 [2.4 to 3.8] | 4.0 [3.3 to 4.8]

3. Secondary Outcome: Core Study Part I: CFB in DAS28 C-reactive Protein (CRP) Score
Description: The DAS28 index is a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, patient global assessment of disease activity score, and CRP value. Total score ranged between 0-10. A DAS28-CRP score of 5.1 or above = high disease activity, a value between 3.2 and 5.1 = moderate disease activity and value between 2.6 and 3.2 = low disease activity, value < 2.6 = disease remission. A positive change in score indicates worsening, and a negative change indicates improvement. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
score on a scale
  Baseline | 5.0 [4.4 to 5.6] | 5.07 [4.4 to 5.7]
  CFB at Week 4: number analyzed (Participants) | 17 | 14
  CFB at Week 4 | 3.4 [2.8 to 4.0] | 4.01 [3.3 to 4.7]
  CFB at Week 8: number analyzed (Participants) | 17 | 13
  CFB at Week 8 | 2.8 [2.2 to 3.4] | 3.81 [3.1 to 4.5]
  CFB at Week 12: number analyzed (Participants) | 17 | 14
  CFB at Week 12 | 3.31 [2.7 to 3.9] | 4.01 [3.3 to 4.7]

4. Secondary Outcome: Core Study Part I: CFB in American College of Rheumatology (ACR) Component: 68 Tender Joint Count (TJC)
Description: The 68 TJC included the 8 distal interphalangeal (IP), 10 proximal IP and 10 metacarpophalangeal (MTP) joints of hands, the 10 MTP and 10 proximal IP joints of feet, the 2 wrists, 2 elbows, 2 shoulders, 2 acromioclavicular, 2 sternoclavicular, 2 temporomandibular, 2 hip, 2 knee, 2 talo-tibial, and 2 mid-tarsal joints. Joint tenderness was graded present (1) or absent (0). Total score is calculated by adding the scores, which range from 0 (no tender joint) to 68 (all tender joints). Lower scores indicate no tender joint and higher scores indicate worsening tender joints. A negative change from Baseline indicates improvement. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: tender joints
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
tender joints
  Baseline | 8.89 [4.9 to 12.9] | 11.18 [7.1 to 15.3]
  CFB at Week 4: number analyzed (Participants) | 18 | 14
  CFB at Week 4 | 5.33 [1.3 to 9.3] | 5.85 [1.5 to 10.2]
  CFB at Week 8: number analyzed (Participants) | 18 | 13
  CFB at Week 8 | 3.72 [-0.3 to 7.7] | 5.1 [0.6 to 9.6]
  CFB at Week 12: number analyzed (Participants) | 17 | 14
  CFB at Week 12 | 4.66 [0.6 to 8.7] | 6.9 [2.6 to 11.2]

5. Secondary Outcome: Core Study Part I: CFB in ACR Component: 66 Swollen Joint Count (SJC)
Description: The 66 SJC included the 8 distal interphalangeal (IP), 10 proximal IP and 10 metacarpophalangeal (MTP) joints of hands, the 10 MTP and 10 proximal IP joints of feet, the 2 wrists, 2 elbows, 2 shoulders, 2 acromioclavicular, 2 sternoclavicular, 2 temporomandibular, 2 knee, 2 talo-tibial, and 2 mid-tarsal joints. Swelling was graded present (1) or absent (0). Total score is calculated by adding the scores, which range from 0 (no swollen joint) to 66 (all swollen joints). Lower scores indicate no swollen joint and higher scores indicate worsening swollen joints. A negative change in Baseline indicates improvement. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: swollen joints
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
swollen joints
  Baseline | 5.78 [3.6 to 7.9] | 8.0 [5.8 to 10.2]
  CFB at Week 4: number analyzed (Participants) | 18 | 14
  CFB at Week 4 | 2.5 [0.4 to 4.6] | 2.5 [0.1 to 4.9]
  CFB at Week 8: number analyzed (Participants) | 18 | 13
  CFB at Week 8 | 1.33 [-0.8 to 3.5] | 2.65 [0.2 to 5]
  CFB at Week 12: number analyzed (Participants) | 17 | 12
  CFB at Week 12 | 2.89 [0.7 to 5.1] | 4.71 [2.4 to 7.0]

6. Secondary Outcome: Core Study Part I: CFB in the 28 TJC
Description: A total of 28 joints were assessed for tenderness. The number of tender joints could range from 0 to 28, where higher values represented more tender joints. The change from Baseline to any time points was averaged among all participants, where negative changes indicated an improvement in disease activity. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: tender joints
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
tender joints
  Baseline | 6.78 [4.6 to 9.0] | 7.24 [5.0 to 9.5]
  CFB at Week 4: number analyzed (Participants) | 18 | 14
  CFB at Week 4 | 3.67 [1.5 to 5.9] | 4.29 [1.9 to 6.7]
  CFB at Week 8: number analyzed (Participants) | 18 | 13
  CFB at Week 8 | 2.39 [0.2 to 4.6] | 3.85 [1.4 to 6.3]
  CFB at Week 12: number analyzed (Participants) | 17 | 14
  CFB at Week 12 | 3.47 [1.2 to 5.7] | 4.43 [2.1 to 6.8]

7. Secondary Outcome: Core Study Part I: CFB in the 28 SJC
Description: A total of 28 joints were assessed for swelling. The number of swollen joints could range from 0 to 28, where higher values represented more swollen joints. The change from Baseline to any time point was averaged among all participants, where negative changes indicated an improvement in disease activity. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: swollen joints
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
swollen joints
  Baseline | 4.97 [3.4 to 6.6] | 6.29 [4.6 to 8.0]
  CFB at Week 4: number analyzed (Participants) | 18 | 14
  CFB at Week 4 | 2.11 [0.5 to 3.7] | 2.47 [0.7 to 4.2]
  CFB at Week 8: number analyzed (Participants) | 18 | 13
  CFB at Week 8 | 0.83 [-0.8 to 2.5] | 2.79 [1.0 to 4.6]
  CFB at Week 12: number analyzed (Participants) | 17 | 14
  CFB at Week 12 | 2.28 [0.6 to 3.9] | 4.51 [2.8 to 6.3]

8. Secondary Outcome: Core Study Part I: CFB in ACR Component: Acute Phase Reactant CRP
Description: A negative change from Baseline in CRP level indicates an improvement. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams per liter (mg/L)
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
milligrams per liter (mg/L)
  Baseline | 45.55 [26.1 to 65.0] | 57.26 [37.3 to 77.2]
  CFB at Week 4: number analyzed (Participants) | 17 | 14
  CFB at Week 4 | 17.53 [-2.1 to 37.1] | 36.74 [15.8 to 57.7]
  CFB at Week 8: number analyzed (Participants) | 18 | 13
  CFB at Week 8 | 14.61 [-4.8 to 34.0] | 32.51 [11.2 to 53.8]
  CFB at Week 12: number analyzed (Participants) | 17 | 14
  CFB at Week 12 | 17.05 [-2.6 to 36.7] | 28.52 [7.0 to 50.0]

9. Secondary Outcome: Core Study Part I: CFB in ACR Component: Acute Phase Reactant ESR
Description: A negative change from Baseline in ESR level indicates an improvement. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeter per hour (mm/h)
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
millimeter per hour (mm/h)
  Baseline | 44.11 [33.8 to 54.4] | 38.82 [28.3 to 49.4]
  CFB at Week 4: number analyzed (Participants) | 16 | 14
  CFB at Week 4 | 24.28 [13.8 to 34.7] | 38.6 [27.5 to 49.7]
  CFB at Week 8: number analyzed (Participants) | 17 | 12
  CFB at Week 8 | 25.4 [15.0 to 35.8] | 25.25 [13.6 to 36.9]
  CFB at Week 12: number analyzed (Participants) | 16 | 14
  CFB at Week 12 | 15.85 [5.3 to 26.4] | 22.41 [10.8 to 34.0]

10. Secondary Outcome: Core Study Part I: CFB in Serum Ferritin Level at Week 12
Description: LS mean was calculated by MMRM analyses.
Time Frame: Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 17 | 14
nanograms per milliliter (ng/mL) | 466.9 [16.0 to 918.0] | 634.71 [170.0 to 1099.0]

11. Secondary Outcome: Core Study Part I: Percentage of Responders With Fever Episodes
Description: Fever is defined as an oral or rectal body temperature greater than 38 degrees Celsius (°C).
Time Frame: Week 12
Population: ITT population included all participants who did not violate any of the following inclusion criteria: diagnosis of adult-onset Still's disease and disease activity based on DAS28 score of ≥ 3.2 at Screening.
Measure: Number; unit: percentage of participants
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
percentage of participants | 8.3 | 0

12. Secondary Outcome: Core Study Part I: CFB in ACR Component: Physician's Global Assessment of Disease Activity Score
Description: The physician's global assessment of disease activity was assessed using a numerical rating scale of 0-10 where 0= no disease activity and 10= activity to maximal disease activity. A negative change from Baseline indicates improvement. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
score on a scale
  Baseline | 5.5 [4.5 to 6.5] | 6.0 [4.9 to 7.1]
  CFB at Week 4: number analyzed (Participants) | 18 | 14
  CFB at Week 4 | 3.06 [2.0 to 4.1] | 3.67 [2.5 to 4.8]
  CFB at Week 8: number analyzed (Participants) | 18 | 13
  CFB at Week 8 | 2.72 [1.7 to 3.8] | 3.56 [2.4 to 4.7]
  CFB at Week 12: number analyzed (Participants) | 17 | 14
  CFB at Week 12 | 2.86 [1.8 to 3.9] | 4.26 [3.1 to 5.4]

13. Secondary Outcome: Core Study Part I: CFB in ACR Component: Participant's Global Assessment of Disease Activity Score
Description: The participant's global assessment of disease activity was assessed using a numerical rating scale of 0-10, where 0= no disease activity and 10= maximal disease activity. A negative change from Baseline indicates improvement. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
score on a scale
  Baseline | 6.08 [4.9 to 7.3] | 5.85 [4.6 to 7.1]
  CFB at Week 4: number analyzed (Participants) | 18 | 14
  CFB at Week 4 | 3.78 [2.6 to 5.0] | 4.74 [3.4 to 6.0]
  CFB at Week 8: number analyzed (Participants) | 17 | 13
  CFB at Week 8 | 2.84 [1.6 to 4.0] | 4.58 [3.2 to 5.9]
  CFB at Week 12: number analyzed (Participants) | 17 | 14
  CFB at Week 12 | 3.63 [2.4 to 4.8] | 4.32 [3.0 to 5.6]

14. Secondary Outcome: Core Study Part I: CFB in ACR Component: Participant's Global Assessment of Pain Score
Description: The participant's global assessment of pain was assessed using a numerical rating scale of 0-10, where 0= no disease activity and 10= maximal disease activity. A negative change from Baseline indicates improvement. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
score on a scale
  Baseline | 6.61 [5.3 to 7.9] | 6.35 [5.0 to 7.7]
  CFB at Week 4: number analyzed (Participants) | 18 | 14
  CFB at Week 4 | 3.61 [2.3 to 4.9] | 4.85 [3.5 to 6.2]
  CFB at Week 8: number analyzed (Participants) | 17 | 13
  CFB at Week 8 | 2.73 [1.4 to 4.0] | 4.18 [2.7 to 5.6]
  CFB at Week 12: number analyzed (Participants) | 17 | 14
  CFB at Week 12 | 3.71 [2.4 to 5.0] | 4.25 [2.8 to 5.7]

15. Secondary Outcome: Core Study Part I: CFB in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: The HAQ measures physical disability and functional status. It has 4 dimensions: disability, pain, drug side effects and dollar costs. The HAQ score is calculated by summing the computed scores for each category and dividing by the number of categories answered. It ranges from 0 (without any difficulty) to 3 (unable to do). A negative change from Baseline indicates improvement. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
score on a scale
  Baseline | 1.31 [0.9 to 1.7] | 1.29 [0.9 to 1.7]
  CFB at Week 12: number analyzed (Participants) | 17 | 14
  CFB at Week 12 | 0.69 [0.3 to 1.1] | 0.98 [0.6 to 1.4]

16. Secondary Outcome: Core Study Part I: Percentage of Responders With American College of Rheumatology Response of 20 (ACR20)
Description: ACR20 response was defined as a ≥ 20% improvement (reduction) compared with Baseline for both 68 TJC and 66 SJC, as well as for three of the additional five ACR core set variables: Participant's Assessment of Pain over the previous 24 hours: using a NRS left end of the line 0=no pain to right end of the line 10=unbearable pain; Participant's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a NRS where left end of the line 0=no disease activity to right end of the line 10=maximum disease activity; HAQ-DI 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant ESR.
Time Frame: Baseline, Week 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
percentage of participants | 61.1 [37.7 to 81.1] | 41.2 [20.1 to 65.0]
Statistical Analysis 1: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 0.3175, Fisher Exact; Difference in Response Rates = 19.9, 95% CI 2-sided [-15.0 to 51.3]

17. Secondary Outcome: Core Study Part I: Percentage of Responders With ACR30
Description: ACR30 response was defined as a ≥ 30% improvement (reduction) compared with Baseline for both 68 TJC and 66 SJC, as well as for three of the additional five ACR core set variables: Participant's Assessment of Pain over the previous 24 hours: using a NRS left end of the line 0=no pain to right end of the line 10=unbearable pain; Participant's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a NRS where left end of the line 0=no disease activity to right end of the line 10=maximum disease activity; HAQ 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant ESR.
Time Frame: Baseline, Week 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
percentage of participants | 61.1 [37.7 to 81.1] | 29.4 [11.7 to 53.7]
Statistical Analysis 1: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 0.0922, Fisher Exact; Difference in Response Rates = 31.7, 95% CI 2-sided [-2.9 to 61.8]

18. Secondary Outcome: Core Study Part I: Percentage of Responders With Modified ACR30
Description: A participant was considered responder if he/she had achieved the incidence of modified adapted response (ACR30 criteria) of at least a 30% improvement in no intermittent fever and had at least 30% improvement in at least 6 of the following 7 measures: tender and swollen 68-joint counts, participant's assessment of pain, participant's global assessment of disease activity, physician's global assessment of disease activity, participant's functional capacity (HAQ-DI score) and acute phase reactant- ESR. Participant were modified ACR30 responders at a given post-randomization visit if they satisfied the modified ACR30 criteria, respectively.
Time Frame: Baseline, Week 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
percentage of participants | 55.6 [32.7 to 76.8] | 23.5 [8.0 to 47.5]
Statistical Analysis 1: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 0.0858, Fisher Exact; Difference in Response Rates = 32.0, 95% CI 2-sided [-1.5 to 61.1]

19. Secondary Outcome: Core Study Part I: Percentage of Responders With ACR50
Description: ACR50 response was defined as a ≥ 50% improvement (reduction) compared with Baseline for both 68 TJC and 66 SJC, as well as for three of the additional five ACR core set variables: Participant's Assessment of Pain over the previous 24 hours: using a NRS left end of the line 0=no pain to right end of the line 10=unbearable pain; Participant's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a NRS where left end of the line 0=no disease activity to right end of the line 10=maximum disease activity; HAQ-DI 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant ESR.
Time Frame: Baseline, Week 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
percentage of participants | 50.0 [27.8 to 72.2] | 17.6 [4.7 to 40.9]
Statistical Analysis 1: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 0.075, Fisher Exact; Difference in Response Rates = 32.4, 95% CI 2-sided [-0.7 to 60.5]

20. Secondary Outcome: Core Study Part I: Percentage of Responders With ACR70
Description: ACR70 response was defined as a ≥ 70% improvement (reduction) compared with Baseline for both 68 TJC and 66 SJC, as well as for three of the additional five ACR core set variables: Participant's Assessment of Pain over the previous 24 hours: using a NRS left end of the line 0=no pain to right end of the line 10=unbearable pain; Participant's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a NRS where left end of the line 0=no disease activity to right end of the line 10=maximum disease activity; HAQ-DI 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant ESR.
Time Frame: Baseline, Week 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
percentage of participants | 27.8 [11.0 to 51.3] | 11.8 [2.0 to 33.7]
Statistical Analysis 1: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 0.4018, Fisher Exact; Difference in Response Rates = 16.0, 95% CI 2-sided [-12.6 to 43.4]

21. Secondary Outcome: Core Study Part I: Percentage of Responders With ACR90
Description: ACR90 response was defined as a ≥ 90% improvement (reduction) compared with Baseline for both 68 TJC and 66 SJC, as well as for three of the additional five ACR core set variables: Participant's Assessment of Pain over the previous 24 hours: using a NRS left end of the line 0=no pain to right end of the line 10=unbearable pain; Participant's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a NRS where left end of the line 0=no disease activity to right end of the line 10=maximum disease activity; HAQ-DI 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant ESR.
Time Frame: Baseline, Week 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
percentage of participants | 11.1 [1.9 to 32.1] | 5.9 [0.3 to 25.8]
Statistical Analysis 1: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 1, Fisher Exact; Difference in Response Rates = 5.2, 95% CI 2-sided [-18.8 to 29.2]

22. Secondary Outcome: Core Study Part I: Percentage of Responders With European League Against Rheumatism (EULAR) Response
Description: EULAR response is based on DAS28-ESR and DAS28-CRP scores. The DAS28 index is a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, subject global assessment of disease activity score, and ESR or CRP value. A DAS28-CRP or ESR score of 5.1 or above = high disease activity, a value between 3.2 and 5.1 = moderate disease activity and value between 2.6 and 3.2 = low disease activity, value < 2.6 = disease remission. EULAR response has 3 categories: EULAR Good response: DAS28 ≤ 3.2 and a change from Baseline < -1.2. EULAR Moderate response: DAS28 >3.2 to ≤ 5.1 or a change from Baseline < -0.6 to ≥ -1.2 or EULAR No response: DAS28 >5.1 or a change from Baseline < -0.6 to ≤ -1.2.
Time Frame: Baseline, Week 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
percentage of participants
  EULAR DAS28-ESR Response | 77.8 [54.7 to 92.5] | 52.9 [29.7 to 75.2]
  EULAR DAS28-CRP Response | 72.2 [48.7 to 89.0] | 47.1 [24.8 to 70.3]
Statistical Analysis 1: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; EULAR DAS28-ESR Response; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 0.1642, Fisher Exact; Difference in Response Rates = 24.8, 95% CI 2-sided [-8.0 to 54.2]
Statistical Analysis 2: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; EULAR DAS28-CRP Response; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 0.1756, Fisher Exact; Difference in Response Rates = 25.2, 95% CI 2-sided [-9.1 to 55.1]

23. Secondary Outcome: Core Study Part I: Percentage of Responders Achieving Low Disease Activity (LDA)
Description: Percentage of responders were defined as the participants who achieved LDA (DAS28 score < 3.2) at Week 12. The DAS28 index is a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, participant global assessment of disease activity score, and ESR or CRP value. Total score ranged between 0-10. A DAS28 score greater than 5.1 implies high disease activity, equal to or less than 3.2 low disease activity, and less than 2.6 remissions.
Time Frame: Week 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
percentage of participants
  DAS28 (ESR) LDA | 33.3 [14.8 to 56.9] | 29.4 [11.7 to 53.7]
  DAS28 (CRP) LDA | 50.0 [27.8 to 72.2] | 23.5 [8.0 to 47.5]
Statistical Analysis 1: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; DAS28 (ESR) LDA; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 1, Fisher Exact; Difference in Response Rates = 3.9, 95% CI 2-sided [-27.7 to 35.0]
Statistical Analysis 2: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; DAS28 (CRP) LDA; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 0.1642, Fisher Exact; Difference in Response Rates = 26.5, 95% CI 2-sided [-6.6 to 56.0]

24. Secondary Outcome: Core Study Part I: Percentage of Responders Achieving Disease Remission and Extended Disease Remission
Description: Participants with disease remission: LDA (DAS28 score< 2.6). The DAS28 index is a composite score of weighted components including both 28 TJC an SJC, participant global assessment of disease activity score, and ESR or CRP value. A DAS28 score greater than 5.1: high disease activity, ≤ 3.2: low disease activity, and less than 2.6: remission. Extended remission criteria included DAS28 < 2.6 and no signs of systemic activity for up to two consecutive study visits till Week 12 defined as any of Yamaguchi´s primary classification criteria for AOSD which included fever attacks at 39 °C for more than a week, arthralgia, salmon red, maculate, urticarial or maculo-papular rash and leukocytosis (white blood cells increase) of > 10000/cubic millimeters (mm^3) with > 80% neutrophils.
Time Frame: Week 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
percentage of participants
  DAS28 (ESR) Remission | 33.3 [14.8 to 56.9] | 11.8 [2.0 to 33.7]
  DAS28 (CRP) Remission | 38.9 [18.9 to 62.3] | 11.8 [2.0 to 33.7]
  Extended Remission | 27.8 [11.0 to 51.3] | 11.8 [2.0 to 33.7]
Statistical Analysis 1: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; DAS28 (ESR) remission; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 0.2285, Fisher Exact; Difference in Response Rates = 21.6, 95% CI 2-sided [-8.1 to 49.9]
Statistical Analysis 2: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; DAS28 (CRP) Remission; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 0.1212, Fisher Exact; Difference in Response Rates = 27.1, 95% CI 2-sided [-4.6 to 54.6]
Statistical Analysis 3: Comparison: Core Study Part I: Canakinumab vs Core Study Part I: Placebo; Extended Remission; Test type: Superiority — Fisher's exact test with a two-tailed level of significance of α = 0.05; p = 0.4018, Fisher Exact; Difference in Response Rates = 16.0, 95% CI 2-sided [-12.6 to 43.4]

25. Secondary Outcome: Core Study Part I: Change in Joint Mobility (Degrees of Motion) Assessed by Neutral Zero Method
Description: Number of joints with limitation of motion according to neutral zero method was assessed which included mobility of joints (elbows, wrists, shoulder joints, hip joints, knee joints, and upper ankle joints) within the reference range/degree. Response is defined as an improvement of ≥ 30%, 50%, 70% and 90% from Baseline. A negative change score indicates improvement. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: degrees
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
degrees
  Baseline | 4.94 [3.0 to 6.9] | 6.29 [4.3 to 8.3]
  Week 12: number analyzed (Participants) | 17 | 14
  Week 12 | 5.37 [3.4 to 7.3] | 6.05 [4.0 to 8.1]

26. Secondary Outcome: Core Study Part I: CFB in Medical Outcome Short Form (SF-36) Health Survey Score
Description: The SF-36 determines overall quality of life assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 contribute to physical component summary score (PCS). Items 5-8 contribute to mental component summary score (MCS). Scores on each item are summed and averaged (range = 0 "worst"-100 "best"). Positive numbers indicate improvement from Baseline. LS mean was calculated by MMRM analyses.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo
Number analyzed (Participants) | 18 | 17
score on a scale
  SF-36 Physical: Baseline | 29.39 [24.5 to 34.3] | 28.73 [23.7 to 33.8]
  SF-36 Physical: CFB at Week 12: number analyzed (Participants) | 17 | 14
  SF-36 Physical: CFB at Week 12 | 41.03 [36.0 to 46.1] | 33.45 [27.9 to 39.0]
  SF-36 Mental: Baseline | 37.8 [32.0 to 43.6] | 46.31 [40.4 to 52.2]
  SF-36 Mental: CFB at Week 12: number analyzed (Participants) | 17 | 14
  SF-36 Mental: CFB at Week 12 | 43.47 [37.6 to 49.3] | 49.82 [43.6 to 56.1]

27. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is an adverse medical event which occurs in a participant of the study and which is not necessarily in a causal relationship with the treatment the participant receives. AEs include symptoms of illnesses, as well as every unfavourable and unintended reaction. SAEs are AEs leading to death, are life-threatening, require hospitalizations or prolongation of hospitalizations, represent an innate malformation or a congenital abnormality.
Time Frame: Up to Month 27
Population: Safety Analysis Set included all participants randomized who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo | Core Study Part II: Canakinumab Responders | Core Study Part II: Placebo Responders | Core Study Part II: Placebo Non-responders | LTE Phase: Canakinumab
Number analyzed (Participants) | 20 | 15 | 14 | 2 | 7 | 7
Participants
  AEs | 16 | 10 | 13 | 2 | 6 | 7
  SAEs | 2 | 0 | 1 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to Month 27
Description: Safety Analysis Set included all participants randomized who received at least one dose of the study drug. 2 participants of the placebo group in Part I received canakinumab at Week 4, as protocol violation, thus, Safety Analysis Set included those additional 2 participants in the canakinumab group.
Arm/Group | Core Study Part I: Canakinumab | Core Study Part I: Placebo | Core Study Part II: Canakinumab Responders | Core Study Part II: Placebo Responders | Core Study Part II: Placebo Non-responders | LTE Phase: Canakinumab
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/15 | 0/14 | 0/2 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/20 | 0/15 | 1/14 | 1/2 | 1/7 | 1/7
Other Adverse Events (participants affected / at risk) | 16/20 | 10/15 | 13/14 | 2/2 | 6/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Study Part I: Canakinumab (N=20) | Core Study Part I: Placebo (N=15) | Core Study Part II: Canakinumab Responders (N=14) | Core Study Part II: Placebo Responders (N=2) | Core Study Part II: Placebo Non-responders (N=7) | LTE Phase: Canakinumab (N=7)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Medical device removal (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Study Part I: Canakinumab (N=20) | Core Study Part I: Placebo (N=15) | Core Study Part II: Canakinumab Responders (N=14) | Core Study Part II: Placebo Responders (N=2) | Core Study Part II: Placebo Non-responders (N=7) | LTE Phase: Canakinumab (N=7)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 2 | 0 | 0 | 3
Injection site rash (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Primary biliary cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infected bite (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 3 | 3 | 0 | 1 | 3
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pertussis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Still's disease (Musculoskeletal and connective tissue disorders) | 5 | 1 | 2 | 1 | 1 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 3 | 1 | 0 | 2 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vulva cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study terminated prior to the planned completion date due to recruitment issues because of the marketing authorization of the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT02204293/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT02204293/SAP_001.pdf